CLINICAL TRIAL: NCT00529243
Title: Virologic Outcomes of Changing Enfuvirtide to Raltegravir in HIV-1 Patients Well Controlled on an Enfuvirtide Based Regimen
Brief Title: Evaluating the Effect of CHanging EnfuvirtidE to Raltegravir in HIV Infected Subjects
Acronym: CHEER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4908
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2011-06-08 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: HIV Infections
Keywords: Treatment Experience; On enfuvirtide
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-0518 (raltegravir) (Experimental): Open label, single arm. All patients to receive MK-0518 400mg orally twice a day for 24 weeks, as substitution for enfuvirtide.
  Interventions: Drug: raltegravir

INTERVENTIONS:
Drug: raltegravir — This is a single-arm, open-label, non-randomized pilot study in human immunodeficiency virus type 1 (HIV-1) positive patients who have an undetectable viral load on their current enfuvirtide containing medication regimen. The treatment regimen will consist of replacing enfuvirtide with MK-0518 400 mg twice a day given as part of the patient's HIV medication regimen. The study regimen will be administered for 24 weeks, with patients given the option of continuing on the study medication past that time if they wish to. Patients serve as their own control as they have viral control (HIV ribonucleic acid (RNA) below limits of quantification) for at least 6 months with enfuvirtide prior to switch to raltegravir.
  Other Names: MK-0518, Isentress

SUMMARY:
The primary objective of this study is:

To assess the virologic effect of changing enfuvirtide to MK-0518(raltegravir) in human immunodeficiency virus type 1(HIV-1) infected patients who have an undetectable level of serum human immunodeficiency virus(HIV) (< 75 copies/ml by branch deoxyribonucleic acid (bDNA) assay, < 50 copies/ml by Ultrasensitive Polymerase Chain Reaction(PCR) assay) on their current HIV medication regimen.

Hypothesis:

HIV-1 infected individuals well controlled on an enfuvirtide containing regimen with HIV RNA levels below limits of quantification can safely have the investigational integrase inhibitor, MK-0518 substituted for enfuvirtide without loss of virologic suppression.

DETAILED DESCRIPTION:
Human immunodeficiency virus type 1(HIV-1) infected patients who have had an undetectable viral load on an enfuvirtide containing regimen at the Kaiser Permanente Hayward, Los Angeles, San Francisco, and Santa Clara Medical Centers will be enrolled. Patients will receive open label MK-0518 (raltegravir) 400mg orally twice a day as substitution for enfuvirtide for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for participation in this study.

  1. Subject is ≥ 18 years of age and able to understand and willing to sign a written informed consent form, which must be obtained prior to initiation of the study.
  2. Documented laboratory diagnosis of HIV-1 infection (positive Enzyme-linked immunosorbent assay (ELISA) HIV-1 antibody test confirmed by western blot, p24 assay, HIV-1 RNA, or culture).
  3. Have documented plasma HIV-1 RNA level(s) of < 75 copies/ml by branched deoxyribonucleic acid(bDNA) assay, or < 50 copies/ml by Ultrasensitive Polymerase Chain Reaction(PCR) for at least 6 months prior to screening visit.
  4. Currently receiving a stable antiretroviral regimen consisting of enfuvirtide plus at least 2 other antiretrovirals for at least 6 months.
  5. Negative serum pregnancy test (females of childbearing potential only) and are willing to use an adequate method of contraception throughout the duration of the study.

Exclusion Criteria:

* Patients who meet any of the following exclusion criteria are not to be enrolled in this study.

  1. Any prior therapy with MK-0518 or any other HIV-1 integrase inhibitor.
  2. Any HIV-1 viral load > 75 copies/ml by bDNA assay, or > 50 copies/ml by Ultrasensitive PCR assay in the 6 months prior to screening visit (A single "blip" of HIV-1 viral load >75 copies but <400 copies by bDNA assay, or >50 copies but <400 copies by Ultrasensitive PCR assay in the six months prior to screening visit with at least one subsequent HIV-1 viral load below the limit of detection will be accepted.)
  3. Any previous known hypersensitivity to components of the study drug formulation.
  4. Weight < 40 kilograms.
  5. Patient requires or is anticipated to require any of the prohibited medications noted in the protocol.
  6. Acute therapy for serious illness (in the opinion of the investigator) within 14 days prior to study entry unless the subject has completed ≥ 7 days of therapy and is considered clinically stable by the investigator.
  7. Any condition which, in the opinion of the investigator, would compromise the subject's ability to participate in the study.
  8. Any active opportunistic infections or Centers for Disease Control and Prevention (CDC) Category C conditions (with the exception of stable cutaneous Kaposi's Sarcoma and wasting syndrome due to HIV infection).
  9. Any malignancy requiring chemotherapy.
  10. Subject has any of the following laboratory results at screening:

      Hemoglobin < 8.0 gr/dl Absolute neutrophil count < 750 cells/ml Platelet count < 40,000 Creatinine > 2.0 or calculated creatinine clearance < 40 ml/min
  11. Female patient who is pregnant or breast-feeding, or expecting to conceive or donate eggs during the study. Male patient who is planning to impregnate or provide sperm donation during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Towner, MD, Principal Investigator — Kaiser Permanente
Locations (8):
- United States (8):
  - Kaiser Anaheim, Anaheim, California
  - Kaiser Hayward, Hayward, California
  - Kaiser Los Angeles, Los Angeles, California
  - Kaiser West Los Angeles, Los Angeles, California
  - Kaiser Panorama City, Panorama City, California
  - Kaiser San Francisco, San Francisco, California
  - Kaiser Santa Clara, Santa Clara, California
  - Kaiser Santa Clarita, Santa Clarita, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multicenter study that enrolled patients from 11 Kaiser Permanente Human Immunodeficiency Virus (HIV) clinics in California. 54 patients were screened. Two patients did not meet protocol inclusion criteria.
Period: Overall Study
Arm/Group | MK-0518 (Raltegravir)
Started | 52
Completed | 49
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Relocated | 1

BASELINE CHARACTERISTICS:
Arm/Group | MK-0518 (Raltegravir)
Number analyzed (Participants) | 52
Age, Continuous [Mean (Full Range); unit: years] | 53 [40 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 48
Region of Enrollment [Number; unit: participants]
  United States | 52
Time of Prior Antiretroviral Therapy Use [Mean (Full Range); unit: years] | 15 [7 to 22]
Number of Past Antiretrovials Used [Mean (Full Range); unit: medications] | 15 [4 to 22]
Time on Enfuvirtide Therapy [Mean (Full Range); unit: days] — mean length of time on enfuvirtide therapy before change to MK-0518 (raltegravir)
  days | 997 [264 to 2457]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Undetectable Human Immunodeficiency Virus (HIV) Viral Load at Week 24.
Description: To assess the virologic effect of changing enfuvirtide to MK-0518 (raltegravir) in human immunodeficiency virus type 1 (HIV-1) infected patients who have an undetectable level of serum HIV (undetectable level of serum HIV defined as < 75 copies/ml by bDNA assay or < 50 copies/ml by Ultrasensitive PCR assay) on their current HIV medication regimen.
Time Frame: 24 Weeks
Population: Analysis used the intent to treat (ITT) population, defined as all patients who received at least one dose of raltegravir.
Measure: Number; unit: participants
Arm/Group | MK-0518 (Raltegravir)
Number analyzed (Participants) | 52
participants | 49

2. Secondary Outcome: Average Change in Cluster of Differentiation 4(CD4) Cell Count From Baseline at Week 24
Description: To study the immunologic effect of changing enfuvirtide to MK-0518 (raltegravir) in HIV-1 infected patients who have an undetectable level of serum HIV (undetectable serum HIV defined as < 75 copies/ml by bDNA assay or < 50 copies/ml by Ultrasensitive PCR assay)on their current HIV medication regimen.
Time Frame: 24 Weeks
Population: Analysis was per intention to treat (ITT) population defined as all patients who received at least one dose of raltegravir.
Measure: Mean (Full Range); unit: cells/mm^3
Arm/Group | MK-0518 (Raltegravir)
Number analyzed (Participants) | 52
cells/mm^3 | 32 [-165 to 1362]

ADVERSE EVENTS:
Time Frame: 33 Weeks
Description: Any adverse event (i.e., a new event or an exacerbation of a pre-existing condition) with an onset date after study drug administration up to the last day on study (including the follow-up, off study medication period of the study), should be recorded.
Arm/Group | MK-0518 (Raltegravir)
Serious Adverse Events (participants affected / at risk) | 3/52
Other Adverse Events (participants affected / at risk) | 12/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0518 (Raltegravir) (N=52)
Septicemia (Blood and lymphatic system disorders) | 1 (1)
Diabetic Ketoacidosis (Endocrine disorders) | 1 (1)
Death (Gastrointestinal disorders) | 1 (1) — Patient with history of gastroparesis & delayed emptying unrelated to his HIV disease died 12 weeks into the study, assessed due to worsening of malnourishment and dehydration not due to his antiretroviral medications or study participation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0518 (Raltegravir) (N=52)
Fatigue (Nervous system disorders) | 3 (3)
alanine aminotransferase (ALT) (Hepatobiliary disorders) | 6 (6)
serum creatinine elevation (Renal and urinary disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
A limitation of our study was the lack of a separate control arm. However, patients did serve as their own control by virtue of at least 6 months of HIV-1 ribonucleic acid(RNA)levels below the level of quantification before enrollment in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes